CLINICAL TRIAL: NCT01709188
Title: The Effects of Musical Dual Task Training on Attention Control and Associated Gait Stability of Patients With Mild to Moderate Dementia
Brief Title: Musical Dual Task Training to Improve Attention Control for Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-2201B; 20216 (Other: University of Kansas)
Record Dates: First submitted 2012-10-01; First posted 2012-10-18 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Dementia
Keywords: Musical Dual Task Training; dementia; attention control; dual task cost; gait stability
MeSH Terms: conditions — Dementia | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Musical Dual Task Training (Experimental): 60 minute individual session once a week across 2 months for a total of 8 sessions.Each session will be led by a qualified music therapist. Within the Musical Dual Task Training session, participant will be asked to sing familiar songs, play simple percussive musical instruments such as paddle drums and shakers, sing while walking, and play instruments while walking.
  Interventions: Behavioral: Musical Dual Task Training
- Walking and Talking (Active Comparator): 60 minute individual session once a week across 2 months for a total of 8 sessions.Each session will be led by a qualified music therapist. Within the walking and talking session, participant will be asked to read a newspaper article prior to a walk and have a conversation with the music therapist based on the content of the news while walking.
  Interventions: Behavioral: Walking and Talking

INTERVENTIONS:
Behavioral: Musical Dual Task Training
  Arms: Musical Dual Task Training
Behavioral: Walking and Talking
  Arms: Walking and Talking

SUMMARY:
The purpose of this project is to determine if the Musical Dual Task Training program improves attention control that influences measures of gait performances under dual tasking, balance, fear of falling, and behavioral disturbance in patients with mild to moderate dementia. This Musical Dual Task Training protocol is structured with musical content and patients are required to do musical tasks including singing and playing instruments contingent on visual or auditory cues while walking. This paradigm is designed to include music making because it involves great demands on attention and memory that might elicit experience-dependent plasticity in the brain. Musical Dual Task Training is proposed to strengthen brain networking for attention control that consequently may improve the gait performances in patients with dementia, as indicated by reducing dual task cost on gait.

ELIGIBILITY:
Inclusion Criteria:

* a mild to moderate dementia diagnosis with Clinical Dementia Rating (CDR) score: .5, 1, or 2
* ability to walk 10 meters independently without the use of a walker or cane, or the assistance by another person

Exclusion Criteria:

* other known neurologic disorders such as stroke or Parkinson's disease
* significant orthopedic, visual, and hearing impairment that hinders ambulation

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the Trail Making Test at 2 months | Baseline and at 2 months
  Trail Making Test Part A requires the participants to draw lines to connect a set of 25 circles as fast as possible following the sequential order of numbers (1,2,3…25) while still maintaining accuracy. Trail Making Test Part B is in a same format, but participants are required to alternates between numbers and letters (1, A, 2, B, etc.). The circles in Part B include both numbers (1 - 13) and letters (A - L). Results for both Part A and Part B are reported as the number of seconds required to complete the task. Higher scores indicate greater impairment.

SECONDARY OUTCOMES:
Change from Baseline on Walking Speed during Dual tasking at 2 Months | Baseline and at 2 months
Change from Baseline on the Timed Up-and-Go test at 2 Months | Baseline and 2 months
Change from Baseline on the 7-item Short Falls Efficacy Scale International at 2 Months | Baseline and at 2 months
Change from Baseline on the Cohen-Mansfield Agitation Inventory scale at 2 months | Baseline and at 2 months
Change from Baseline on Stride Lengths during Dual Tasking at 2 Months | Baseline and at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Pei, MD, PhD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Medical Foundation, Taoyuan District, Taiwan, Taiwan

REFERENCES:
- [Derived] van der Steen JT, van der Wouden JC, Methley AM, Smaling HJA, Vink AC, Bruinsma MS. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2025 Mar 7;3(3):CD003477. doi: 10.1002/14651858.CD003477.pub5. PMID 40049590